CLINICAL TRIAL: NCT06283095
Title: Management of Obstructive Sleep Apnea Syndrome by Expansion Palatoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ET Zarief (Other)
Responsible Party: Sponsor-Investigator, ET Zarief, Principle investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSA
Record Dates: First submitted 2023-11-14; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): we will do expansion palatoplasty
  Interventions: Procedure: expansion palatoplasty

INTERVENTIONS:
Procedure: expansion palatoplasty — surgical procedure

SUMMARY:
The study will be conducted to evaluate the outcome of expansion palatoplasty in management of OSAS.

DETAILED DESCRIPTION:
Expansion palatopladty will be conducted on patients with obstructive sleep apnea patients to evaluate the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* Body mass index < 30 kg/m2 (weight /height in m2)
* Mild to moderate OSAS
* Sagittal collapse of the lateral pharyngeal walls proved by Drug induced sleep endoscopy (DISE).

Exclusion Criteria:

* • Refusing enrollment into the study.

  * Pregnant women.
  * Refusing the surgery
  * Contraindication to anaesthesia
  * Patients with multilevel of obstruction.
  * Serious psychiatric, neurological and cardiopulmonary (COPD or corpulmonale) diseases.
  * Uncorrected hypothyroidism.
  * Severe OSAS.
  * Craniofacial anamolies.
  * Central& mixed apnea
  * Morbid obesity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation the outcome of expansion palatoplasty in management of OSAS. | Six months
  Polysomngrophy

SECONDARY OUTCOMES:
Expansion palatoplasty in Obstructive sleep apnea patients | Six months
  Drug induced sleep endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Enas T Zarief, Principal Investigator — Assuit U
Locations (1):
- ASSUIT, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Managment of OSAS
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Three years
Access Criteria: OSAS
URL: http://enas.tharwat23@gmail.com